CLINICAL TRIAL: NCT07109427
Title: Impact of an Electronic Health Record Maintenance Alert on PSA Screening Rates in a 10-Hospital Integrated Health System
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 202507064
Record Dates: First submitted 2025-07-31; First posted 2025-08-07 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Prostate Cancer; Cancer of the Prostate
Keywords: PSA Screening; Clinically Significant Prostate Cancer; African American men; Electronic Health Record
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Annual PSA Health Maintenance Reminder (Experimental): An annual health maintenance reminder will be implemented for all men who meet the American Cancer Society guidelines for average- and high-risk eligibility criteria. The goal is to encourage their primary care provider (PCP) to engage in a shared decision-making discussion with the patient about the benefits and risks of prostate cancer screening.
  This alert will appear in the health maintenance reminder section of the electronic health record (EHR).
  Although all providers with access to EPIC can view the alert, it is typically the PCPs who review and take action on alerts in the health maintenance reminder section.
  Interventions: Other: Annual PSA Health Maintenance Reminder

INTERVENTIONS:
Other: Annual PSA Health Maintenance Reminder — The annual health maintenance reminder does not mandate PSA screening for eligible patients. Instead, it recommends that primary care providers (PCPs) initiate a shared decision-making discussion with their patients. As part of this conversation, patients will be informed of their individual risk factors-including race, family history, and germline mutations-and can then make an informed choice about whether to proceed with PSA screening.

SUMMARY:
- The investigators propose a clinical trial to evaluate the impact of annual shared decision making for PSA screening, supported by system-level enhancements to promote evidence-based care:

* Defined referral thresholds within the health maintenance reminder, aligned with clinical risk stratification per NCCN guidelines.
* Enhanced clinical decision support (CDS) tools to reduce provider variation and ensure guideline-concordant screening and referral practices.
* The goal is to reduce late-stage presentation without increasing overdiagnosis-ensuring that prostate cancer screening is both accessible and clinically effective.

ELIGIBILITY:
Eligibility Criteria:

* Receive care within the BJC Health System
* Have had at least one primary care physician appointment in the calendar year of PSA screening (primary care)
* Be male
* Not have a history of prostate cancer
* Meet one of the following risk criteria:

  * High Risk for Prostate Cancer

    * African American, between the ages of 40 and 75 (inclusive), or
    * Family history of prostate, breast, ovarian, and/or pancreatic cancer, or
    * Known familial germline mutation OR
  * Average Risk for Prostate Cancer

    * Between the ages of 50 and 75 (inclusive)

Ages: 40 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40000 (Estimated)
Dates: Start 2025-08-11 (Actual); Primary Completion 2031-08-31 (Estimated); Study Completion 2031-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in PSA screening completion rates in the BJC East Health System | Through 5 years
  The overall PSA screening rate will be calculated as the number of PSA screening tests that are ordered by PCPs who will receive the alert and completed by patients within a year of the ordering date, divided by the total number of eligible patients.

SECONDARY OUTCOMES:
Proportion of men diagnosed with clinically significant prostate cancer (Gleason score ≥ 7) | Through 5 years
Incidence of advanced and metastatic disease at diagnosis of prostate cancer | Through 5 years
Incidence of early-stage prostate cancer | Through 5 years
Stage distribution of prostate cancer diagnoses | Through 5 years
Biopsy rates | Through 5 years
Percent of PSA screening ordered but not completed | Through 5 years
Median PSA at time of diagnosis | Through 5 years
Evaluate the agreement between 3T MRI and biomarker test results | Through 5 years
  The 3T MRI and biomarker tests are used to help determine whether a biopsy is necessary. The investigators will categorize the results as positive versus negative and the agreement will be gauged based on Kappa coefficient.
PSA screening rate by age group | Through 5 years
  Age groups will include 40-49, 50-70, and 70-75
PSA screening rate by race | Through 5 years
PSA screening rate by comorbidity burden | Through 5 years
PSA screening rate by insurance coverage | Through 5 years
PSA screening rate by provider | Through 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Lannis Hall, M.D., MPH, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu